CLINICAL TRIAL: NCT03336268
Title: Project POINT: Effectiveness and Scalability of an Overdose Survivor Intervention
Acronym: POINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alan McGuire, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1706859955; R33DA045850 (NIH)
Record Dates: First submitted 2017-10-26; First posted 2017-11-08 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Substance Use Disorders; Overdose
Keywords: Opioid Use Disorder; Peer Recovery Coach
MeSH Terms: conditions — Substance-Related Disorders; Drug Overdose; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POINT (Experimental): This arm will be offered both POINT services (in addition to standard emergency care) and enrollment in study data collection. If they choose to enroll in POINT, they may choose whether or not to enroll in data collection, as it is not required. Should they enroll in data collection, they will be consented and enrolled in the research study as a participant in the POINT study arm.
  Interventions: Behavioral: POINT
- Standard Care (No Intervention): This arm will only be offered enrollment in study data collection, as they will receive standard emergency care. If they choose to enroll, they will be consented in the research study as the Standard Care arm.

INTERVENTIONS:
Behavioral: POINT — A recovery coach meets patients in the ED after they have been revived from an overdose to offer a range of services including an assessment of high-risk behaviors, Hep C/HIV testing, harm reduction counseling, and treatment referrals with follow-up to either a medication for opioid use disorder (MOUD) provider, detoxification services, or an inpatient treatment setting. Patients are offered a take-home naloxone kit and assistance with Medicaid enrollment. Close collaboration with the local community mental health provider ensures POINT patients have their first assessment for MOUD within 1-2 business days of ED discharge. Also, recovery coaches offer to accompany patients to intake appointments or criminal justice and child welfare meetings as part of the standard care they deliver.
  Arms: POINT

SUMMARY:
The investigators seek to assess the effectiveness of Project POINT (Planned Outreach, Intervention, Naloxone, and Treatment). As originated in Indianapolis, Project POINT is a collaboration between Indianapolis Emergency Medical Services (EMS), the Eskenazi Emergency Department, Midtown Mental Health, and researchers at Indiana University. POINT is a quality improvement initiative that connects trained outreach workers with emergency department (ED) patients who experienced a non-fatal overdose. A member of the POINT team (a recovery coach or care coordinator with specialized training) meets patients after they have experienced an opioid overdose and, following a model of patient-centered care, offers them a range of evidence-based services including a brief assessment of high-risk behaviors, Hepatitis C and HIV testing, harm reduction counseling informed by motivational interviewing, and treatment referrals with follow-up to either a medication for opioid use disorder (MOUD) provider, detoxification services, or an inpatient treatment setting

The primary goal of this project is the establishment of POINT as an effective and scalable intervention for engaging patients in MAT. This study employs a Hybrid Type 1 effectiveness implementation design to take full advantage of current POINT expansion efforts currently happening in Indiana. The goal of this study is to replicate POINT in new hospitals and test its feasibility through (a) assessment of the chosen implementation strategy and (b) the testing of research protocols and secondary data collection procedures.

DETAILED DESCRIPTION:
STUDY DESIGN The investigators will conduct the pilot study at Indiana University Health Methodist Hospital in Indianapolis, Indiana and at Indiana University Health Ball Memorial Hospital in Muncie, Indiana.

The pilot study includes two study arms.

Arm(1): Regarding the POINT intervention, a recovery coach (someone certified by the Indiana Counselors' Association on Alcohol and Drug Abuse to deliver recovery supports who has lived experience with addiction) meets patients in the ED after they have been revived from an overdose (patients are typically alert and oriented, as the overdoes reversal drug completely stops the effect of opioids in their system, and patients will not be approached until a physician has determined they are eligible for release). As part of the POINT program, the recovery coach offers the patient a range of evidence-based services including a brief assessment of high-risk behaviors, Hepatitis C and HIV testing, harm reduction counseling informed by motivational interviewing, and treatment referrals with follow-up to either a medication for opioid use disorder (MOUD) provider, detoxification services, or an inpatient treatment setting-with most patients choosing MOUD referral. Patients are offered a take-home naloxone kit (the overdose reversing drug, which is offered as part care delivered by the recovery coach) and assistance with Medicaid enrollment. Close collaboration with the local community mental health provider ensures POINT patients have their first assessment for MOUD within 1-2 business days of ED discharge. Grounded in the concept of critical time intervention, recovery coaches provide over the phone or in person support to navigate barriers to care throughout the recovery process. Also as part of the POINT program, recovery coaches offer to accompany patients to intake appointments or criminal justice and child welfare meetings as part of the standard care they deliver (no data collection for research purposes will occur as part of this service provision). The entire care transition process takes between 2 weeks and several months, and POINT leaves the door open so patients can re-engage at any point they require help overcoming recovery barriers.

Arm (2): The standard care arm will consist of basic referral to services by informing patients of available treatment options in the community.

RANDOMIZATION & ENROLLMENT For each day of the study, researchers will randomly select during which of the shifts patients will enroll into the POINT arm and which will enroll into standard care (morning shift (8am-3:59pm), evening (4pm-11:59pm), and overnight (12am-7:59am). Any individual who is discharged from the ED for an opioid overdose or for an opioid-related health issue, including opioid withdrawal, abscess (from IV drug use) or active opioid intoxication will be eligible for the study. The research team and recovery coaches will receive an electronic alert from emergency medical services any time an overdose patient is admitted to the ED. A recovery coach will be sent to the ED on POINT shifts, and a research assistant will be sent on non-POINT shifts. Once they have confirmed that the admit is reason is either an opioid overdose or an opioid-related issue, they will read the questions on the DSM-5 for Opioid Use Disorder screening tool. Any individual who is at least 18 years of age and is discharged from the ED for an overdose an opioid related health issue AND scores at least a "1" on the opioid use disorder screening tool will be initially eligible for the study; they must also be cleared for discharge and medically stable and capable of providing consent. Depending on the arm of the study patients are being recruited to on that shift, either the recovery coach or the research assistant will inform the patient of the study and request their consent to participate.

Researchers will not fully disclose the purposes of the research to the standard care arm because (1) Methodist Hospital and Ball Memorial were planning on implementing POINT outside of the context of this study and because their ability to staff recovery coaches is limited anyway, we are not creating any disparity in patients ability to access point that would not naturally exist and (2) we are concerned that full disclosure of the purposes would unnecessarily upset standard care patients who might desire the services after learning of them.

The study site plans to implement Project POINT regardless of the research study. Therefore, all recovery coach duties are part of POINT prescribed services that would be carried out regardless of the research. The investigators are randomizing the shift during which POINT is delivered to take advantage of the fact that they are not able to fully staff all hospital shifts with a recovery coach--thus allowing us to test the intervention's effectiveness. Only those patients in the standard care arm will be asked to complete data collection activities that would not be completed outside of the research study.

After study consent, all subjects will be asked to complete a structured interview with either a recovery coach (POINT group) or a research assistant (standard care). This interview will occur in the ED, and it can take between 30-60 minutes and covers the following topics: demographics, social support; living arrangements, drug use, context of current overdose, treatment history, interest in recovery services, use of strategies to reduce risks related to drug use, HIV and Hepatitis C, physical and mental health, adverse childhood experiences, and detailed contact information. Additionally, the RA or recovery coach will collect detailed contact information on the participant to increase chances of being able to follow up with the participant. This contact information will be entered into a separate database and will not be linked to questionnaire responses.

The investigators will also collect information from the following existing secondary data sources:

* Indiana Network for Patient Care (contains hospital and overdose admission data)
* INSPECT (contains prescription information for controlled substances)
* Division of Mental Health and Addiction (contains methadone treatment information)
* Indiana Office of Medicaid Planning and Policy (contains Medicaid enrollment information)
* Indiana Department of Child Services (contains child welfare involvement information)
* Valle Vista Health System (contains addiction and mental health treatment data)
* Midtown Community Mental Health (contains mental health treatment data)
* Clean Slate (contains addiction treatment data)

As part of the POINT project, recovery coaches engage with POINT patients for two weeks (reaching out to patients every 2-3 days until the patient is successfully engaged in recovery services), but this may last longer (several months) depending on patient need and desire for continued assistance. Recovery coaches will not be collecting data for study purposes during this time; rather, any information they collect will be their employment purposes as a recovery coach. Standard care patients are not seen after the initial referral.

The investigators will also collect data from hospital records and government and public health databases on patients enrolled in the study after obtaining a release for these information from subjects. The investigators will collect methadone data from the Division of Mental Health and Addiction (DMHA), prescribing information related to controlled substances from INSPECT (prescription drug monitoring system), the hospital admission data from Indiana Network for Patient Care (INPC), overdose death information form coroner records, insurance information from Medicaid, child welfare system involvement form the Department of Child Services (DCS), and publicly available criminal justice data. A third party, Regenstrief Institute, will work with all of these systems to securely obtain and merge the data and to de-identify the data before sharing it with the research team.

ELIGIBILITY:
Inclusion Criteria:

1. Revived from a drug overdose or admitted to the ED for an opioid-related health issue, including opioid withdrawal, abscess (from IV opioid use), endocarditis (from IV opioid use), or active opioid intoxication
2. Score at least "1" on the DSM-5 for Opioid Use Disorder screening tool
3. Eligible for discharge from the Methodist or Ball Memorial Hospital Emergency Department and deemed able to speak to research staff by ED staff
4. Be 18 or older
5. Be medically stable (i.e., cleared to leave the ED by a physician) and capable of providing consent.

Exclusion Criteria:

(a) Unable to answer the 3 study competency questions that indicate capability of providing consent.

(Individuals discharged from the ED during a POINT shift who do not wish to participate in the study are still eligible to receive POINT services.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Watson, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watson DP, Tillson M, Taylor L, Xu H, Ouyang F, Beaudoin FL, O'Donnell D, McGuire AB. Results From the POINT Pragmatic Randomized Trial: An Emergency Department-Based Peer Support Specialist Intervention to Increase Opioid Use Disorder Treatment Linkage and Reduce Recurrent Overdose. Subst Use Addctn J. 2024 Jul;45(3):378-389. doi: 10.1177/29767342231221054. Epub 2024 Jan 9. PMID 38258819

RESULTS

PARTICIPANT FLOW:
Groups:
- POINT: This arm will be offered both POINT services (in addition to standard emergency care) and enrollment in study data collection. If they choose to enroll in POINT, they may choose whether or not to enroll in data collection, as it is not required. Should they enroll in data collection, they will be consented and enrolled in the research study as a participant in the POINT study arm.
  POINT: A recovery coach meets patients in the ED after they have been revived from an overdose to offer a range of services including an assessment of high-risk behaviors, Hep C/HIV testing, harm reduction counseling, and treatment referrals with follow-up to either a medication assisted treatment (MAT) provider, detoxification services, or an inpatient treatment setting. Patients are offered a take-home naloxone kit and assistance with Medicaid enrollment. Close collaboration with the local community mental health provider ensures POINT patients have their first assessment for MAT within 1-2 business days of ED discharge. Also, recovery coaches offer to accompany patients to intake appointments or criminal justice and child welfare meetings as part of the standard care they deliver.
Period: Overall Study
Arm/Group | POINT | Standard Care
Started | 159 | 90
Completed | 159 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 249 participants enrolled in the study, only 243 were included in the analysis (POINT arm=157; Standard Care arm=86).
  A total of 6 participants, including 2 participants from the POINT arm and 4 participants from the Standard Care arm, were excluded from the analysis because they were unable to be matched to administrative records.
Groups:
- Total: Total of all reporting groups
Arm/Group | POINT | Standard Care | Total
Number analyzed (Participants) | 157 | 86 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.1) | 37.2 (11.7) | 35.8 (10.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 68 | 32 | 100
  Male | 88 | 54 | 142
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 153 | 84 | 237
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 11 | 28
  White | 139 | 75 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 157 | 86 | 243
Insurance Status [Count of Participants; unit: Participants]
  Healthy Indiana Plan (HIP) | 91 | 45 | 136
  Medicaid | 17 | 8 | 25
  Medicare | 7 | 6 | 13
  Private (exchange, employer-based) | 10 | 3 | 13
  Other | 1 | 4 | 5
  None | 30 | 20 | 50
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Opioid Overdose
Description: Total participants presenting to the emergency department (ED) for an opioid overdose.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 18 | 9
  Within 6 months pre-enrollment | 10 | 6
  Within 3 months pre-enrollment | 5 | 4
  Within 1 month pre-enrollment | 0 | 3
  Within 1 month post-enrollment | 3 | 3
  Within 3 months post-enrollment | 11 | 6
  Within 6 months post-enrollment | 15 | 11
  Within 12 months post-enrollment | 26 | 15

2. Secondary Outcome: Medication for Opioid Use Disorder (MOUD) Engagement
Description: Total participants with buprenorphine prescriptions, naltrexone prescriptions, or dosed methadone.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 46 | 16
  Within 6 months pre-enrollment | 36 | 9
  Within 3 months pre-enrollment | 24 | 7
  Within 1 month pre-enrollment | 8 | 3
  Within 1 month post-enrollment | 36 | 14
  Within 3 months post-enrollment | 49 | 26
  Within 6 months post-enrollment | 65 | 28
  Within 12 months post-enrollment | 77 | 38

3. Secondary Outcome: Duration of Medication for Opioid Use Disorder (MOUD) Engagement
Description: Total days of supply of buprenorphine prescriptions, naltrexone prescriptions, or methadone dosed for participants with a medication for opioid use disorder (MOUD).
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Population: Of the 243 participants matched to administrative records, only 243 unique participants were found to have a prescription for a MOUD within the outcome measure time frame and included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
days
  Within 12 months pre-enrollment: number analyzed (Participants) | 46 | 16
  Within 12 months pre-enrollment | 45.0 [16.0 to 194.0] | 44.6 [27.0 to 121.0]
  Within 6 months pre-enrollment: number analyzed (Participants) | 36 | 9
  Within 6 months pre-enrollment | 41.0 [14.0 to 88.1] | 29.0 [18.0 to 97.0]
  Within 3 months pre-enrollment: number analyzed (Participants) | 24 | 7
  Within 3 months pre-enrollment | 16.0 [10.4 to 43.4] | 36.9 [14.0 to 48.9]
  Within 1 month pre-enrollment: number analyzed (Participants) | 8 | 3
  Within 1 month pre-enrollment | 14.0 [9.0 to 19.0] | 14.0 [9.0 to 14.0]
  Within 1 month post-enrollment: number analyzed (Participants) | 36 | 14
  Within 1 month post-enrollment | 17.7 [6.7 to 24.9] | 15.9 [8.0 to 30.0]
  Within 3 months post-enrollment: number analyzed (Participants) | 49 | 26
  Within 3 months post-enrollment | 39.0 [21.0 to 64.3] | 30.0 [8.0 to 63.3]
  Within 6 months post-enrollment: number analyzed (Participants) | 65 | 28
  Within 6 months post-enrollment | 47.6 [21.6 to 95.0] | 47.3 [36.0 to 106.5]
  Within 12 months post-enrollment: number analyzed (Participants) | 77 | 38
  Within 12 months post-enrollment | 84.0 [30.0 to 168.0] | 53.5 [22.0 to 207.3]

4. Secondary Outcome: Emergency Department Presentations
Description: Total participants presented to the Emergency Department for any medical reason.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 99 | 52
  Within 6 months pre-enrollment | 77 | 43
  Within 3 months pre-enrollment | 55 | 30
  Within 1 month pre-enrollment | 29 | 18
  Within 1 month post-enrollment | 34 | 18
  Within 3 months post-enrollment | 63 | 30
  Within 6 months post-enrollment | 82 | 47
  Within 12 months post-enrollment | 102 | 56

5. Secondary Outcome: Inpatient Hospital Admissions
Description: Total participants admitted to the hospital for any medical reason.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 44 | 23
  Within 6 months pre-enrollment | 29 | 17
  Within 3 months pre-enrollment | 21 | 9
  Within 1 month pre-enrollment | 10 | 4
  Within 1 month post-enrollment | 48 | 17
  Within 3 months post-enrollment | 52 | 20
  Within 6 months post-enrollment | 58 | 27
  Within 12 months post-enrollment | 71 | 36

6. Secondary Outcome: Time to Relapse
Description: Relapse-free survival probability for 6 months and 12 months. Participants who did not have ED presentation were censored at 1) time of 6 month or 12 months, 2) one's last day in the study, 3) overdose death date, whichever is the earliest.
Time Frame: Enrollment through 6 & 12 months post-enrollment
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
probability
  Within 6 months post-enrollment | 0.85 [0.79 to 0.90] | 0.84 [0.75 to 0.91]
  Within 12 months post-enrollment | 0.77 [0.70 to 0.83] | 0.74 [0.63 to 0.82]

7. Secondary Outcome: Medicaid Enrollment for Participants Without Insurance
Description: Total participants without insurance coverage at enrollment that enrolled in Medicaid.
Time Frame: Enrollment through 3 months, 6 months, and 12 months post-enrollment
Population: Only participants without insurance at the time of enrollment (N=50) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 30 | 20
Participants
  Within 3 months post-enrollment | 10 | 7
  Within 6 months post-enrollment | 13 | 8
  Within 12 months post-enrollment | 16 | 15

8. Secondary Outcome: Child Welfare Involvement
Description: Total open child welfare cases.
Time Frame: 3 years pre-enrollment through 1 year post-enrollment
Measure: Number; unit: open cases
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
open cases
  36 months pre-enrollment | 20 | 13
  24 months pre-enrollment | 19 | 12
  12 months pre-enrollment | 10 | 8
  6 months pre-enrollment | 5 | 4
  3 months pre-enrollment | 2 | 1
  1 month pre-enrollment | 0 | 0
  1 month post-enrollment | 1 | 1
  3 months post-enrollment | 1 | 2
  6 months post-enrollment | 4 | 4
  12 months post-enrollment | 9 | 4

9. Secondary Outcome: Incarceration
Description: Total days experienced incarceration.
Time Frame: 3 years pre-enrollment through 1 year post-enrollment
Population: Though enrollment occurred in two Indiana counties, incarceration records were only accessible for the 212 participants enrolled in Marion County (129 in the POINT arm and 83 in Standard Care) as the other county does not have publicly accessible records. Of these, a total of 145 unique participants were found to have been incarcerated within the outcome measure time frame and included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 83 | 62
days
  Within 3 years pre-enrollment | 88.0 [17.0 to 263.0] | 73.5 [11.0 to 347.0]
  Within 2 years pre-enrollment: number analyzed (Participants) | 78 | 56
  Within 2 years pre-enrollment | 39.0 [11.0 to 157.0] | 30.5 [9.0 to 183.5]
  Within 12 months pre-enrollment: number analyzed (Participants) | 51 | 35
  Within 12 months pre-enrollment | 10.0 [3.0 to 47.0] | 18.0 [5.0 to 76.0]
  Within 6 months pre-enrollment: number analyzed (Participants) | 32 | 26
  Within 6 months pre-enrollment | 6.5 [3.0 to 21.5] | 10.5 [5.0 to 71.0]
  Within 3 months pre-enrollment: number analyzed (Participants) | 20 | 22
  Within 3 months pre-enrollment | 5.5 [2.5 to 19.5] | 8.5 [4.0 to 25.0]
  Within 1 month pre-enrollment: number analyzed (Participants) | 12 | 9
  Within 1 month pre-enrollment | 6.5 [3.5 to 14.5] | 3.0 [2.0 to 13.0]
  Within 1 month post-enrollment: number analyzed (Participants) | 15 | 10
  Within 1 month post-enrollment | 13.0 [5.0 to 24.0] | 5.5 [3.0 to 8.0]
  Within 3 months post-enrollment: number analyzed (Participants) | 29 | 19
  Within 3 months post-enrollment | 11.0 [4.0 to 44.0] | 9.0 [4.0 to 50.0]
  Within 6 months post-enrollment: number analyzed (Participants) | 44 | 29
  Within 6 months post-enrollment | 15.0 [4.5 to 51.0] | 10.0 [3.0 to 39.0]
  Within 12 months post-enrollment: number analyzed (Participants) | 53 | 37
  Within 12 months post-enrollment | 19.0 [5.0 to 104.0] | 13.0 [6.0 to 47.0]

10. Post Hoc Outcome: Opioid Prescriptions (Excluding Medications for Opioid Use Disorder (MOUD) Prescriptions)
Description: Total participants with opioid prescriptions, excluding Medications for Opioid Use Disorder (MOUD) prescriptions.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 44 | 30
  Within 6 months pre-enrollment | 31 | 20
  Within 3 months pre-enrollment | 18 | 15
  Within 1 month pre-enrollment | 18 | 15
  Within 1 month post-enrollment | 18 | 15
  Within 3 months post-enrollment | 8 | 6
  Within 6 months post-enrollment | 14 | 7
  Within 12 months post-enrollment | 19 | 9

11. Post Hoc Outcome: Benzodiazepine Prescriptions
Description: Total participants with benzodiazepine prescriptions.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 17 | 11
  Within 6 months pre-enrollment | 16 | 8
  Within 3 months pre-enrollment | 13 | 6
  Within 1 month pre-enrollment | 6 | 5
  Within 1 month post-enrollment | 10 | 5
  Within 3 months post-enrollment | 15 | 6
  Within 6 months post-enrollment | 17 | 7
  Within 12 months post-enrollment | 21 | 11

12. Post Hoc Outcome: Narcan Prescriptions
Description: Total participants with Narcan prescriptions.
Time Frame: 1 year pre-enrollment through 1 year post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 157 | 86
Participants
  Within 12 months pre-enrollment | 10 | 4
  Within 6 months pre-enrollment | 7 | 3
  Within 3 months pre-enrollment | 5 | 3
  Within 1 month pre-enrollment | 3 | 0
  Within 1 month post-enrollment | 7 | 3
  Within 3 months post-enrollment | 11 | 3
  Within 6 months post-enrollment | 13 | 6
  Within 12 months post-enrollment | 17 | 9

13. Post Hoc Outcome: Medicaid Enrollment for Participants With Insurance
Description: Total participants with insurance coverage at enrollment that enrolled in Medicaid.
Time Frame: Enrollment through 3 months, 6 months, and 12 months post-enrollment.
Population: Only participants with insurance at the time of enrollment (N=193) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | POINT | Standard Care
Number analyzed (Participants) | 127 | 66
Participants
  Within 3 months post-enrollment | 78 | 38
  Within 6 months post-enrollment | 83 | 41
  Within 12 months post-enrollment | 86 | 47

ADVERSE EVENTS:
Time Frame: One year pre-enrollment through one year post-enrollment.
Description: Serious adverse events included: all-cause mortality, opioid-related overdoses, presentation to the emergency department for any medical reason, and admission to the hospital for any medical reason. Data for these events come from administrative data pulls.
  Adverse events included: violation of confidentiality, discomfort due to the interview process, and disclosure of information about harm to self or others. Information for these events come from direct participant reporting.
Arm/Group | POINT | Standard Care
All-Cause Mortality (participants affected / at risk) | 25/157 | 16/86
Serious Adverse Events (participants affected / at risk) | 102/157 | 56/86
Other Adverse Events (participants affected / at risk) | 0/157 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POINT (N=157) | Standard Care (N=86)
Opioid Overdose (Injury, poisoning and procedural complications) | 29 | 19 — Opioid overdoses, including deaths caused by opioid-related poisonings and presentations to the emergency department for opioid-related overdoses.
Emergency Department Presentation (General disorders) | 102 | 56 — Presentation to the emergency department for any medical reason.
Inpatient Hospital Admission (General disorders) | 71 | 36 — Inpatient hospital admissions for any medical reason.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POINT (N=157) | Standard Care (N=86)
Violation of Confidentiality (Social circumstances) | 0 | 0
Discomfort Due to Interview (Social circumstances) | 0 | 0
Disclosure of Information About Harm to Self/Others (Social circumstances) | 0 | 0

LIMITATIONS AND CAVEATS:
Because of IRB requirements, the control arm was enrolled by research assistants and the treatment arm was enrolled by peers. Higher treatment arm enrollment was likely due to peers' relationship building role. The COVID pandemic stopped quality improvement efforts and enrollment before the issue could be full addressed. Thus, the study was unable to address enrollment discrepancies or reach the target sample (n=712). The study was likely underpowered to detect change in the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT03336268/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT03336268/ICF_001.pdf